CLINICAL TRIAL: NCT01936584
Title: Validation of Quality of Life Assessment After Laparoscopic TAPP and TEP Surgery of Inguinal Hernias Using EuraHS of Life Score and Carolinas Comfort Scale™
Acronym: LIQUOR
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2013/381
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Primary Unilateral Inguinal Hernias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TAPP repair: TAPP repair for inguinal hernia
  Interventions: Procedure: TAPP repair for inguinal hernias; Other: EuraHS-QoL questionnaire; Other: Carolina Comfort Scale
- TEP repair: TEP repair for inguinal hernia
  Interventions: Procedure: TEP repair for inguinal hernia; Other: EuraHS-QoL questionnaire; Other: Carolina Comfort Scale

INTERVENTIONS:
Procedure: TAPP repair for inguinal hernias
  Groups: TAPP repair
Procedure: TEP repair for inguinal hernia
  Groups: TEP repair
Other: EuraHS-QoL questionnaire — questionnaire administration
Other: Carolina Comfort Scale — questionnaire administration

SUMMARY:
A multicenter observational study trial validating Quality of Life assessment using EuraHS Quality of Life score and Carolinas Comfort scale™ in patients before and after laparoscopic unilateral inguinal hernia repair.

Depending on the treating physician patients will receive a TAPP or TEP repair for their inguinal hernia and a self-gripping mesh will be used for the repair (Parietex Progrip Mesh).

Primary endpoint will be assessment by the EuraHS-QoL at 1 year after laparoscopic repair of an unilateral inguinal hernia using the Anatomic ProGrip™ Laparoscopic self-fixating mesh.

Secondary endpoints are assessment of the QoL 3 preoperative, 3 weeks and 1 year postoperative, recurrence rate at 12 months, intra-operative and post-operative complications, post-operative hospital stay, operation time and time to place the mesh, VAS (Visual Analog Scale) for pain at several control points, VRS (Verbal Rating Score) for pain at 3 weeks and 12 months, pain medication needed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient or his/her legal representative
* Primary unilateral inguinal hernia undergoing a preperitoneal laparoscopic repair.

Exclusion Criteria:

* No written informed consent
* Recurrent groin hernia
* Open hernia repair
* Bilateral hernias
* Concomitant repair of another abdominal hernia eg umbilical hernia
* Hernia repair combined with another surgical procedure
* Emergency operations, like incarcerated hernias
* Patients under the age of 18 years and over 80 years
* Pregnant women
* ASA score 4 or more
* Patients unable to perform the QoL assessment, because of language barrier or intellectual incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing laparoscopic unilateral inguinal hernia repair
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
assessment of the EuraHS-QoL | 1 year after start study
  questionnaire assessment

SECONDARY OUTCOMES:
change in EuraHS-QoL assessment | preoperatively (at inclusion), 3 weeks and 1 year, postoperatively recurrence rate at 12months
  clinical evaluation, Carolina Comfort Scale™ questionnaire, EuraHS-QoL questionnaire, Visual Analogue Scale and Verbal Rating Score.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - AZ Maria Middelares, Ghent
  - University Hospital Ghent, Ghent
  - Heilig Hart Ziekenhuis, Mol

REFERENCES:
- [Derived] Muysoms FE, Vanlander A, Ceulemans R, Kyle-Leinhase I, Michiels M, Jacobs I, Pletinckx P, Berrevoet F. A prospective, multicenter, observational study on quality of life after laparoscopic inguinal hernia repair with ProGrip laparoscopic, self-fixating mesh according to the European Registry for Abdominal Wall Hernias Quality of Life Instrument. Surgery. 2016 Nov;160(5):1344-1357. doi: 10.1016/j.surg.2016.04.026. Epub 2016 Jun 14. PMID 27316825